CLINICAL TRIAL: NCT01809275
Title: A Phase 1/2 Randomized, Placebo-Controlled, Double-Blind Study of the Induction of Clinical Response and Remission by QBECO in Subjects With Moderate to Severe Crohn's Disease
Brief Title: Safety and Treatment Effect of QBECO in Moderate to Severe Crohn's Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Qu Biologics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: QBECO-01
Record Dates: First submitted 2013-03-08; First posted 2013-03-12 (Estimated); Last update posted 2016-08-23 (Estimated); Status verified 2016-08

CONDITIONS: Crohn's Disease; Inflammatory Bowel Disease
Keywords: Crohn's Disease; Inflammatory Bowel Disease; CDAI
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- QBECO (Experimental): Individualized maintenance dose ranging from 0.01 - 0.2 mL, administered subcutaneously, every other day for a maximum of 16 weeks
  Interventions: Drug: QBECO
- Placebo (Placebo Comparator): Individualized maintenance dose ranging from 0.01 - 0.2 mL, administered subcutaneously, every other day for a maximum of 16 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: QBECO
  Arms: QBECO
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety profile and to obtain an indication as to the therapeutic effect of QBECO induction treatment on clinical improvement in moderate to severe Crohn's Disease.

ELIGIBILITY:
Inclusion Criteria:

* An adult, age 18 and above
* Diagnosed with Crohn's disease AT LEAST six (6) months prior to screening
* Crohn's disease diagnosis was verified by one of these procedures: 1) Colonoscopy 2) Capsule endoscopy 3) Computed Tomography (CT) scan 4) Magnetic Resonance Imaging (MRI) 5) Ultrasound
* Active Crohn's disease at the time of screening
* Female participants: Agree to practice two effective methods of contraception, at the same time, from the time of signing the informed consent form, during the entire study treatment and for two (2) months after taking the last dose of study treatment.
* Male participants: Agree to practice effective barrier contraception during the entire study treatment period and for two (2) months after taking the last dose of study treatment.

Exclusion Criteria:

* Currently pregnant or breastfeeding
* Have known or suspected hypersensitivity to any component of the product
* Had more than three (3) small bowel resections or diagnosis of short bowel syndrome
* Currently anticipate undergoing any major surgical intervention for Crohn's disease during the next six (6) months
* Previously been treated with any Qu Biologics' Site Specific Immunomodulators (SSIs) for any disease
* Diagnosed with chronic (i.e., long term) hepatitis B or C infection
* Diagnosed with congenital (i.e., existing at or before birth) or acquired immunodeficiency (i.e., lack of body defense system). For example, human immunodeficiency virus (HIV) infection, organ transplantation (i.e., specifically received an organ from a donor), etc.
* Daily use of narcotic drugs containing opiates (such as morphine, codeine, etc.) for pain control
* Have a current or recent history (within the past 12 months) of alcohol dependence or illicit drug use, with the exception of medicinal marijuana prescribed by a physician
* Have a history of cancer within the last five (5) years. Exceptions may apply for cervical cancer and some forms of skin cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2013-03; Primary Completion 2016-02 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Safety | 8 weeks
  Assessing adverse events, concomitant therapies, clinical chemistry, hematology, urinalysis chemistry
Clinical improvement | 8 weeks
  Assessing the change in Crohn's Disease Activity Index (CDAI) from baseline

SECONDARY OUTCOMES:
Clinical remission | 8 weeks
  Assessing the change in Crohn's Disease Activity Index (CDAI) from baseline
Clinical response | 8 weeks
  Assessing the change in Crohn's Disease Activity Index (CDAI) from baseline
Intestinal inflammation | 8 weeks
  Assessing the change in fecal calprotectin from baseline
Systemic inflammation | 8 weeks
  Assessing the change in C-reactive protein (CRP) from baseline

CONTACTS AND LOCATIONS:
Overall Officials: M D, Study Director — Qu Biologics Inc.; M D, Principal Investigator — GI Research Institute
Locations (4):
- Canada (4):
  - University of Calgary, Calgary, Alberta
  - University of Alberta Zeidler Ledcor Centre, Edmonton, Alberta
  - GI Research Institute, Vancouver, British Columbia
  - Toronto Digestive Disease Associates, Vaughan, Ontario

REFERENCES:
- [Derived] Sutcliffe S, Kalyan S, Pankovich J, Chen JMH, Gluck R, Thompson D, Bosiljcic M, Bazett M, Fedorak RN, Panaccione R, Axler J, Marshall JK, Mullins DW, Kabakchiev B, McGovern DPB, Jang J, Coldman A, Vandermeirsch G, Bressler B, Gunn H. Novel Microbial-Based Immunotherapy Approach for Crohn's Disease. Front Med (Lausanne). 2019 Jul 19;6:170. doi: 10.3389/fmed.2019.00170. eCollection 2019. PMID 31380382
- See also: Informational website for this trial — http://www.quibd.com